CLINICAL TRIAL: NCT03851016
Title: The Effectiveness of Life Story Book on Depression and Meaning in Life for Mentally Alert Residents of Nursing Homes
Brief Title: Life Story Book With Mentally Alert Residents of Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Theresa C. Chrisman, Theresa C. Chrisman, PhD., LMSW, University of Houston
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Study00001439
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Depressive Symptoms; Quality of Life
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A switching replication design was employed to examine the effects of the Life Story Book (LSB). Two comparable nursing homes were allocated to each intervention. Participants in each nursing home received the same intervention at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life Story Book Intervention First, Then Usual Care (Experimental): Participants first received the Life Story Book Intervention once a week for 3 weeks. After a washout period of 1 week, they then received the Usual Care Intervention for 3 weeks. Posttests were then conducted for 1 week.
  Interventions: Behavioral: Life Story Book
- Usual Care First, Then Life Story Book Intervention (Experimental): Participants first received the Usual Care Intervention for 3 weeks. After a washout period of 1 week, they then received the Life Story Book Intervention once a week for 3 weeks. Posttests were then conducted for 1 week.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Life Story Book — Life story Book is intended to allow a person the opportunity to reminisce chronologically through their life and capture their life stories into a book.
  Arms: Life Story Book Intervention First, Then Usual Care
Behavioral: Usual Care — Three weeks of Usual Care with no visits from research team
  Arms: Usual Care First, Then Life Story Book Intervention

SUMMARY:
The objective of this study is to study the effects of the Life Story Book intervention on depressive symptoms and meaning in life for mentally alert residents of nursing homes.

DETAILED DESCRIPTION:
Two nursing homes were recruited to participate. One nursing home will receive the Life Story Book intervention while the other half receives Usual Care intervention. The interventions were then switched, and the participants who received Usual Care intervention received the Life Story Book intervention while the home that received Life Story Book intervention received Usual Care intervention. The study consisted of two treatment periods of 3 weeks separated by a washout period of 1 week.

Life Story Book provides a person with the opportunity to chronologically share their life experiences and memories. This three-1 hour reminiscence intervention is designed to provide a person with the opportunity to review their past and capture their life story into something tangible. The Life Story Book includes a combination of written information, photographs of significant people, places or events, and personal narratives from the stages of life that the person would like to include.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak English
* A resident of the nursing home
* A score of 4 or higher on the Six-Item Screener

Exclusion Criteria:

* A score of 4 or higher on the Six-item Screener

Min Age: 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa C Chrisman, LMSW, Principal Investigator — University of Houston; Allen Rubin, PhD, Study Chair — University of Houston
Locations (2):
- United States (2):
  - Sharpview Residence and Rehabilitation Center, Houston, Texas
  - Cambridge Health Rehab Center, Richmond, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKeown J, Clarke A, Ingleton C, Ryan T, Repper J. The use of life story work with people with dementia to enhance person-centred care. Int J Older People Nurs. 2010 Jun;5(2):148-58. doi: 10.1111/j.1748-3743.2010.00219.x. PMID 20925716
- [Background] McKeown J, Clarke A, Repper J. Life story work in health and social care: systematic literature review. J Adv Nurs. 2006 Jul;55(2):237-47. doi: 10.1111/j.1365-2648.2006.03897.x. PMID 16866815
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Sutcliffe C, Cordingley L, Burns A, Mozley CG, Bagley H, Huxley P, Challis D. A new version of the geriatric depression scale for nursing and residential home populations: the geriatric depression scale (residential) (GDS-12R). Int Psychogeriatr. 2000 Jun;12(2):173-81. doi: 10.1017/s104161020000630x. PMID 10937538
- [Background] Steger, M. F., Frazier, P., Oishi, S., & Kaler, M. The meaning in life questionnaire: Assessing the presence of and search for meaning in life. Journal of counseling psychology 53(1): 80-93, 2006.
- [Background] Gibson, F. Reminiscence and life story work: A practice guide. Jessica Kingsley Publishers, 2011.
- [Background] Haight, Barbara K., and Barrett S. Haight. The handbook of structured life review. Baltimore, MD: Health Professions Press, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 residents were screened for eligibility between April 08, 2019 and April 12, 2019 from two comparable nursing homes in the Houston Texas Metropolitan area.
Pre-assignment Details: 24 of the 27 participants, 12 from each home met inclusion criteria. The two nursing homes were allocated by the PI to either Life Story Book Intervention first or Usual Care first. All participants in the same nursing home received the same intervention at the same time.
Groups:
- Life Story Book Intervention First, Then Usual Care: Participants first received the Life Story Book Intervention for one hour each week for 3 weeks. After a washout period of 1 week and measures collected (Time 2), they then received the Usual Care intervention for 3 weeks. Posttests (Time 3) were conducted the week after the Usual Care intervention.
- Usual Care First, Then Life Story Book Intervention: Participants first received the Usual Care Intervention for 3 weeks. After a washout period of 1 week and measures collected (Time 2), they then received the Life Story Book Intervention for one hour a week for 3 weeks. Posttests (Time 3) were conducted the week after the Life Story Book Intervention.
Period: First Intervention (3 Weeks)
Arm/Group | Life Story Book Intervention First, Then Usual Care | Usual Care First, Then Life Story Book Intervention
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Washout (1 Week)
Arm/Group | Life Story Book Intervention First, Then Usual Care | Usual Care First, Then Life Story Book Intervention
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Life Story Book Intervention First, Then Usual Care | Usual Care First, Then Life Story Book Intervention
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Life Story Book Intervention First, Then Usual Care: Participants first received the Life Story Book Intervention for one hour a week for three weeks. After a washout period of 1 week, they then received three weeks of usual care.
- Usual Care First, Then Life Story Book Intervention: Participants received three weeks of usual care first. After a washout period of 1 week, they then received three weeks of the Life Story Book Intervention
- Total: Total of all reporting groups
Arm/Group | Life Story Book Intervention First, Then Usual Care | Usual Care First, Then Life Story Book Intervention | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.1 (11) | 72.1 (11.7) | 74.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 6 | 5 | 11
  Ethnicity: African American | 3 | 4 | 7
  Ethnicity: Asian | 2 | 0 | 2
  Ethnicity: Hispanic | 0 | 1 | 1
Education, Categorical [Count of Participants; unit: Participants]
  Grades 9-11 | 2 | 1 | 3
  High School or GED | 4 | 2 | 6
  Some College/Tech | 2 | 7 | 9
  College Graduate, plus | 3 | 0 | 3
Marital Status, Categorical [Count of Participants; unit: Participants]
  Widow (R) | 7 | 4 | 11
  Divorced | 3 | 3 | 6
  Single | 1 | 2 | 3
  Married | 0 | 1 | 1
Length of Time at Residence [Count of Participants; unit: Participants]
  Less than 1 Year | 5 | 1 | 6
  One-two years | 6 | 6 | 12
  Three or more years | 0 | 3 | 3
Katz Index of Independence in Activities of Daily Living (ADL) Continuous [Mean (Standard Deviation); unit: units on a scale] — The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment. 6 = High (patient independent) 0 = Low (patient very dependent).
  The mean score and standard deviation for each nursing home (A and B) was calculated to compare the physical functioning ability of each home's participants.
  units on a scale | 1.27 (.65) | 3.0 (2.3) | 2.135 (1.8)
Religion [Count of Participants; unit: Participants]
  Protestant | 8 | 8 | 16
  Catholic/Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Scores for Geriatric Depression Scale at 3 Weeks
Description: The Geriatric Depression Scale (Residential) (GDS-12R) is a validated, self-reported instrument assessing depression over the past 7 days. It is a "yes/no" format. Possible scores range from 0 (no depressive symptoms) to 10 (depression). A score of 0 to 4 is normal; scores ≥ 4 are significant for depressive symptoms; scores ≥ 08 is almost always indicative of depression. A score ≥ 5 points should warrant a follow-up comprehensive assessment.
Time Frame: Baseline and 3 weeks
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Life Story Book Intervention: Participants who received the Life Story Book intervention in either the first three weeks or the last three weeks of the study.
- Usual Care: Participants who received Usual Care in either the first or last 3 weeks of the study.
Arm/Group | Life Story Book Intervention | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | 1.00 (2.07) | -.29 (1.68)
Statistical Analysis 1: Comparison: Life Story Book Intervention vs Usual Care; Null hypothesis is that there would be no difference in change of depressive symptoms between Life Story Book Intervention and Usual Care. A multivariate analysis of covariance (MANCOVA) models with the GDS-12R at baseline as the covariate, and the treatment group and study site as factors. The test was performed with a significance level of 0.05. A sample size of 20 was needed to provide 90% power to detect a 5 point difference in depressive symptoms; Test type: Superiority; p = .113, Mancova

2. Primary Outcome: Change From Baseline in Mean Scores for Meaning in Life Questionnaire Sub-Scale Presence of Meaning (POM) at 3 Weeks.
Description: Meaning in Life was measured using the Meaning in Life Questionnaire (MLQ), created by Steger et al. The MLQ has two sub-scales which assess the presence of meaning (POM) (how much a person feels their life has meaning) and the search for meaning (how much a person strives to find meaning and understanding in their life). The two sub-scale measures, which consist of 10 items on a 7-point Likert scale, range from 1-absolutely true to 7-absolutely untrue: five items for presence of meaning (POM) and five items for search for meaning (SFM).
  A POM score > 24 indicates the person feels their life has meaning and purpose.
Time Frame: Baseline and 3 weeks
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Life Story Book Intervention | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | .952 (6.18) | -13.10 (13.78)
Statistical Analysis 1: Comparison: Life Story Book Intervention vs Usual Care; Null hypothesis is that there would be no difference in change of Presence of Meaning (POM) between Life Story Book Intervention and Usual Care. A multivariate analysis of covariance (MANCOVA) models with the POM at baseline as the covariate, and the treatment group and study site as factors. The test was performed with a significance level of 0.05. A sample size of 20 was needed to provide 90% power to detect a 5 point difference in POM; Test type: Superiority; p = .123, Mancova

3. Primary Outcome: Change From Baseline in Mean Scores for Meaning in Life Questionnaire Sub-Scale Search for Meaning (SFM) at 3 Weeks
Description: Meaning in Life was measured using the Meaning in Life Questionnaire (MLQ), created by Steger et al.The MLQ has two sub-scales which assess the presence of meaning (how much a person feels their life has meaning) and the search for meaning (how much a person strives to find meaning and understanding in their life). The two sub-scale measures, which consist of 10 items on a 7-point Likert scale, range from 1-absolutely true to 7-absolutely untrue: five items for presence of meaning (POM) and five items for search for meaning (SFM).
  An SFM score of < 24 indicates the person is not seeking meaning in their life.
Time Frame: Baseline and 3 weeks
Population: All participants who received each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Life Story Book Intervention | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale | -2.62 (10.11) | 12.24 (13.11)
Statistical Analysis 1: Comparison: Life Story Book Intervention vs Usual Care; The null hypothesis is that there would be no difference in change of Search for Meaning (SFM) between Life Story Book Intervention and Usual Care. A multivariate analysis of covariance (MANCOVA) models with the SFM at baseline as the covariate, and the treatment group and study site as factors. The test was performed with a significance level of 0.05. A sample size of 20 was needed to provide 90% power to detect a 5 point difference in SFM; Test type: Superiority; p = .910, Mancova

ADVERSE EVENTS:
Time Frame: Through the study completion, an average of 9 weeks, no serious or other adverse effects were observed.
Groups:
- Life Story Book Intervention: Two comparable nursing homes (NH) were allocated to either Life Story Book Intervention first (NH-A) or Usual Care first (NH-B) Participants in the same NH will receive the same intervention.
- Usual Care Intervention: Two comparable nursing homes (NH) were randomly allocated to either Life Story Book Intervention first (NH-A) or Usual Care first (NH-B) Participants in the same NH will receive the same intervention.
Arm/Group | Life Story Book Intervention | Usual Care Intervention
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03851016/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03851016/Prot_SAP_001.pdf